CLINICAL TRIAL: NCT05039216
Title: Biobank for Inflammatory Chronic Diseases and Osteoporosis of TOULouse
Brief Title: Biobank for Inflammatory Chronic Diseases and Osteoporosis
Acronym: BIOTOUL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0163
Record Dates: First submitted 2021-09-06; First posted 2021-09-09 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Spondyloarthritis; Osteoporosis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylarthritis; Osteoporosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients initiating a biotherapy or a target treatment: Blood sampling
  Interventions: Biological: Blood sampling
- patients with chronic inflammatory rheumatism, weakening osteopathy or mechanical pathology: Blood sampling
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — 4 tubes of 7 mL will be sampled

SUMMARY:
The aim of this study is to constitute a biobank for patients followed in the Rheumatology center of Toulouse University Hospital for a chronic inflammatory rheumatism including rheumatoid arthritis (RA), spondyloarthritis(SpA), and psoriatic arthritis (PsA) or a chronic bone disease including osteoporosis in order to identify biomarkers associated with therapeutic response.

DETAILED DESCRIPTION:
Biologic ant targeted synthetic disease modifying anti-rheumatic drugs (bDMARDs and tsDMARDs) have greatly improved the prognosis of chronic inflammatory diseases. To date, many bDMARDs and tsDMARDs targeting different immunologic mechanisms are available to treat RA, SpA or PsA. However, the choice of the treatment and its mechanism of action is based on physician decision and experience. Indeed, predictive clinical and biological factors associated with therapeutic response that could help the physician to make his/her choice are lacking. The aim of BIOTOUL is to collect and store biologic samples in patients with RA, SpA or PsA who begin a new bDMARD or tsDMARD. This biobank will permit to study several biomarkers and assess the association between such markers and response to therapy.

Furthermore, osteoporosis is a chronic disease leading to fractures and disability. Several ant-osteoporotic drugs are now available and biomarker(s) that would help the physician to choose the best therapeutic sequence are lacking. BIOTOUL will also include patients with osteoporosis to identify biomarkers associated with severity and response to anti-osteoporotic treatments.

ELIGIBILITY:
Inclusion Criteria:

* Chronic inflammatory rheumatism including RA, SpA or PsA or patients with primary or secondary osteoporosis
* With National Health Assurance
* Able to consent to the study

Exclusion Criteria:

* Pregnancy or breastfeeding
* Not able to give a consent
* Severe anemia (Hb<10g/L)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: monocentric observational longitudinal study
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2026-09-02 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
EULAR response after 3 months | after 3 months
  EULAR response after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Adeline RUYSSEN-WITRAND, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Purpan University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No